CLINICAL TRIAL: NCT00639132
Title: The Natural History of Metachromatic Leukodystrophy
Acronym: NH-US
Status: Withdrawn | Type: Observational
Why Stopped: Merged with a broader study of rare diseases once moved to Pittsburgh
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Maria Escolar, Professor, University of Pittsburgh
Other Study IDs: NH-US
Record Dates: First submitted 2008-03-11; First posted 2008-03-19 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Metachromatic Leukodystrophy
Keywords: Natural History; Metachromatic Leukodystrophy; Disease Progression
MeSH Terms: conditions — Leukodystrophy, Metachromatic; Disease Progression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, CSF and urine

SUMMARY:
There have not been longitudinal studies which track patients' neurologically or developmentally in a systematic manner. By simultaneously tracking patients' neurodevelopment along with neuroimaging and neurophysiologic studies it becomes much easier to draw conclusions on the differential effects of the disease process and any available treatments that patients might receive. In addition, many of the gene mutations, which cause MLD have not been linked to the age of onset or the expected disease course.

DETAILED DESCRIPTION:
Metachromatic leukodystrophy (MLD), an autosomal recessively inherited lysosomal storage disorder, causes a deficiency of arylsulfatase A. This results in accumulation of sulfated glycolipids (sulphatide) within lysosomes of myelin forming cells in the central and peripheral nervous system and to a lesser extent in lysosomes of cells comprising the liver, kidneys, and gallbladder. The disease is characterized by progressive demyelination with wide variability in clinical onset and severity. Depending upon the age at onset and disease progression, MLD may be classified as late infantile (6 months to 4 years), early juvenile (4 to 6 years), late juvenile (6 to 16 years), and adult (>16 years). In the late infantile and early juvenile forms, blindness, gait disturbances, loss of speech, loss of hearing, and quadriparesis are common signs. In older children and adults the disease may present with gait disturbances, mental regression, and behavioral abnormalities. Disease progression, also variable, results in death within a few years to several decades; however, disease progression among affected siblings seems to follow a similar course, unlike many other leukodystrophies.

Bone marrow transplantation (BMT) has been the only partially effective treatment reported for MLD. BMT has been shown to halt disease progression when asymptomatic patients achieve engraftment prior to the age at which symptoms occurred in an affected, symptomatic sibling. Despite stabilization of the clinical course when receiving BMT before symptoms, patients' neurophysiologic test abnormalities persist. The clinical implication of this finding has not been further researched. Patients who show mild to moderate progression of their disease prior to transplantation continue to exhibit disease progression to severe impairment. However, specific degrees of clinical impairment in neurodevelopmental function have not been monitored to determine what level of cognitive and motor impairment can be present and still allow the patient to confer benefits from treatment. Patients with late infantile MLD appear to benefit the least from the transplantation process based on preliminary unpublished data. Several case report studies for patients with late infantile MLD indicate delayed, but continued progression of the disease despite BMT, while others suggest initial deterioration followed by stabilization.

Transplantation with allogenic hematopoietic stem cells has been shown to positively influence the disease progression of other lysosomal storage diseases such as Hurler Syndrome and Krabbe Disease and testing for enzyme replacement for MLD is already underway. For future researchers to be able compare the benefits of children with MLD who receive treatment to those who remained untreated, a better understanding of the natural progression of late infantile MLD is necessary. The current literature contains studies of individual or small groups of MLD patients that tracked intelligence quotients and neurophysiologic function, but did not correlate this with patients' neurodevelopment. A longitudinal study of a larger population of patients with late infantile MLD has yet to be performed. This protocol is a longitudinal observational study to capture natural history data in patients with late infantile MLD. This data will provide baseline neurobehavioral, neuroimaging, and neurophysiological information that can in the future be used to evaluate treatment effects.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have a confirmed diagnosis of MLD as defined by:

   ASA activity < 10 nmol/h/mg in leukocytes

   Presence of elevated sulfatide in urine
2. The patient must have voluntary function (as judged by the investigator), including cognitive and motor function that is no more than 3 standard deviations below normal at the time of enrollment.
3. The patient must have an age at the time of screening birth to < 6 years
4. The patient must have had onset of symptoms before the age of 4 years
5. The subject and his/her guardian(s) must have the ability to comply with the clinical protocol

Exclusion Criteria:

1. Known multiple sulfatase deficiency
2. Presence of major congenital abnormality
3. Presence of known chromosomal abnormality and other neurological conditions unrelated to MLD that can affect psychomotor development
4. History of hematopoietic stem cell transplantation
5. Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical condition
6. Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the principal investigator, would preclude participation in the trial
7. Use of any investigational product within 30 days prior to study enrollment or currently enrolled in another study which involves clinical investigations.
8. The patient's parent(s) and/or legal guardian is unable to understand the nature, scope, and possible consequences of the study.
9. Patient is unable to comply with the protocol, i.e. inability to return for follow-up evaluations or otherwise unlikely to complete the study as determined by the principal investigator.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with biochemical evidence of MLD including low levels of arylsulphatase A white cell activity and increased amounts of urinary sulphatide excretion are eligible for the study. A total of 10 patients representing various ranges of disease severity are expected to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-03-11 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Results of cognitive and motor testing | baseline, 6 months, 12 months and then yearly
  Patients receive standardized neurodevelopmental testing Cognitive Motor Language

SECONDARY OUTCOMES:
Audiology | baseline, 6, 12, then yearly
  Audiologic examination
MRI | yearly
  Magnetic Resonance Imaging of the Brain